CLINICAL TRIAL: NCT01324258
Title: A Phase I Trial of GSK1120212 and GSK1120212 in Combination With Gemcitabine in Japanese Subjects With Solid Tumors
Brief Title: Trial of GSK1120212 and GSK1120212 in Combination With GEM in Japanese Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114784
Record Dates: First submitted 2011-01-22; First posted 2011-03-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: pancreatic cancer (combination with gemcitabine); Non-small cell lung cancer (combination with gemcitabine); solid tumors (single agent); MEK inhibitor; GSK1120212; biliary cancer (combination with gemcitabine); urothelial cancer (combination with gemcitabine)
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms | interventions — trametinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1120212 (Experimental): Part 1-Dose escalation will be conducted to assess PK after single dosing and safety, tolerability, PK and efficacy of GSK1120212 in Japanese subjects with solid tumors using a continuous daily dosing schedule.
  Interventions: Drug: GSK1120212; Drug: Gemcitabine
- GSK1120212+Gemcitabine (Experimental): Part 2-Further evaluate the safety, tolerability, PK, and efficacy of GSK1120212 in combination with gemcitabine in subjects with non-small cell lung cancer, pancreatic cancer, biliary cancer, urothelial cancer or other tumor types for which 4-week schedule of gemcitabine has been approved using the recommended dose from Part 1 (single agent).
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: GSK1120212 — Part1 and Part2
  Arms: GSK1120212
Drug: Gemcitabine — Part2

SUMMARY:
This is the first clinical experience in Japan with GSK1120212, a novel MEK inhibitor. This study is designed to identify recommended doses and regimens in Japanese subjects for the future development of GSK1120212.

DETAILED DESCRIPTION:
GSK1120212 has demonstrated anti-proliferative activity against a broad range of tumors cell lines and xenograft models. To date, MEK inhibitors have demonstrated evidence of both pharmacodynamic and clinical activity in early trials.

This is the first clinical experience in Japan with GSK1120212, a novel MEK inhibitor. This study is designed to identify recommended doses and regimens in Japanese subjects for the future development of GSK1120212.

This study will be conducted in subject with solid tumors, and GSK1120212 single agent treatment to assess safety, tolerability, PK and efficacy (Part 1) and combination treatment with gemcitabine in subjects with non-small cell lung cancer, pancreatic cancer, biliary cancer, urothelial cancer or other tumor types for which gemcitabine has been approved in 4-week schedule to assess safety, tolerability, PK and efficacy(Part 2) will be conducted in the same protocol.

ELIGIBILITY:
Inclusion Criteria:

Correspond Part 1 (Single agent) and Part 2 (Combination)

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Age 20 years old or older at consent given
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Negative for hepatitis B surface (HBs) antigen, hepatitis virus Bc (HBc) antibody, and HBs antibody. HBs antigen-negative subjects who test positive for both HBc antibody and HBs antibody or either of them may be eligible when their HBV DNA quantification result is negative
* Negative HCV antibody test
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the time of the first dose of GSK1120212 until 16 weeks after the last dose of GSK1120212
* A female subject is eligible to participate if she is of;Non-childbearing potential females or female subjects with child-bearing potential must agree to use contraception until four weeks after the last dose of GSK1120212 to sufficiently minimize the risk of pregnancy at that point

Part 1 -Dose escalation single agent part

* Histologically or cytologically confirmed diagnosis of solid tumor malignancy that is not responsive to standard therapies or for which there is no approved or curative therapy. Subjects with primary brain tumor are excluded
* Adequate organ system functions as defined below; Absolute neutrophil count≥1,200/uL Hemoglobin≥9g/dL Platelets≥75,000/uL PT/INR and APTT≤1.3xULN Albumin≥2.5g/dL Total bilirubin≤1.5xULN AST and ALT≤2.5xULN Creatinine≤ULN OR Calculated creatinine clearance≥50mL/min OR 24-hour urine creatinine clearance≥50mL/min Left ventricular Ejection fraction≥LLN by ECHO or MUGA

Part 2 -Combination part

* Tumor type criteria;Histologically or cytologically confirmed diagnosis of solid tumor malignancy. Eligible are the cancers for which gemcitabine has been approved in 4-week schedule;1,000mg/m2 weekly for 3weeks followed by 1 week rest at the 4th week, including non-small cell lung cancer, pancreatic cancer, biliary cancer, and urothelial cancer, to which gemcitabine monotherapy is considered to be appropriate
* Adequate organ system functions as defined below; Absolute neutrophil count≥1,500/uL Hemoglobin≥9g/dL Platelets≥100,000/uL PT/INR and APTT1≤1.3xULN Albumin≥2.5g/dL Total bilirubin≤1.5xULN AST and ALT≤2.5xULN Creatinine≤ULN OR Calculated creatinine clearance≥50mL/min OR 24-hour urine creatinine clearance≥50mL/min Left ventricular Ejection fraction≥LLN by ECHO or MUGA

Exclusion Criteria:

Correspond Part 1 (Single agent) and Part 2 (Combination)

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter preceding the first dose of GSK1120212. Or use of an other investigational drug within 28 days or five half-lives, whichever is longer preceding the first dose of GSK1120212
* Previous treatment with a MEK inhibitor
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or subinvestigator, contraindicates their participation
* History of interstitial lung disease or pneumonitis
* Current use of a prohibited medication
* Any major surgery, radiotherapy, or immunotherapy within 21 days before initiation of GSK1120212. Or chemotherapy regimens with delayed toxicity within 21 days before initiation of GSK1120212. Or chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the two weeks before initiation of GSK1120212
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* QTc B≥480 msecs
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks
* History or evidence of current≥Class II congestive heart failure as defined by New York Heart Association
* History or evidence of current clinically significant uncontrolled arrhythmias
* History of HIV infection
* Evidence of severe or uncontrolled systemic diseases
* Unresolved toxicity greater than CTCAE (Version 3.0) Grade 1 from previous anti-cancer therapy except alopecia
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to dimethyl sulfoxide (DMSO)
* Pregnant or lactating female
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol
* Unwillingness or inability to follow the procedures outlined in the protocol

Part 1 -Dose escalation single agent part

* History of another malignancy
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs

Part 2 -Combination part

* History of another malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2013-07-08 (Actual); Study Completion 2013-07-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Until a subject has a Dose Limiting Toxicity, withdraws from the study or dies

SECONDARY OUTCOMES:
To assess pharmacokinetics (PK) parameter (AUC, Cmax, tmax etc.) values for GSK1120212 | Cycle0, Cycle1 Day1,8,15,22, Cycle2 Day1 in Part 1
  Individual subject parameter values as well as a descriptive summary (mean, standard deviation, median, minimum, maximum, geometric mean, and the standard deviation, CV% and 95% confidence interval of log-transformed parameters) by dose cohort will be reported.
To assess pharmacokinetics (PK) parameter (AUC, Cmax, tmax, etc.) values for GSK1120212 and Gemcitabine | Cycle1 Day15 in Part2
  Individual subject parameter values as well as a descriptive summary (mean, standard deviation, median, minimum, maximum, geometric mean, and the standard deviation, CV% and 95% confidence interval of log-transformed parameters) by dose cohort will be reported.
Number of participants with the indicated tumor response defined by RECIST v1.1 | Every eight weeks during the study
Serum level of cyctokines | Cycle1 Day15 in Part1 and Part2
Tissue level of expression of the indicated protein including pERK and Ki67 if possible | Cycle1 Day15 in Part1 and Part2
Tissue level of gene mutation including BRAF and KRAS if possible | Cycle1 Day15 in Part1 and Part2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Kasuga A, Nakagawa K, Nagashima F, Shimizu T, Naruge D, Nishina S, Kitamura H, Kurata T, Takasu A, Fujisaka Y, Okamoto W, Nishimura Y, Mukaiyama A, Matsushita H, Furuse J. A phase I/Ib study of trametinib (GSK1120212) alone and in combination with gemcitabine in Japanese patients with advanced solid tumors. Invest New Drugs. 2015 Oct;33(5):1058-67. doi: 10.1007/s10637-015-0270-2. Epub 2015 Aug 12. PMID 26259955
- See also: Results for study 114784 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114784?search=study&search_terms=114784#rs